CLINICAL TRIAL: NCT01945424
Title: Sanofi Pasteur Quadrivalent Influenza Vaccine Pregnancy Registry Protocol
Brief Title: Sanofi Pasteur Quadrivalent Influenza Vaccine (QIV) Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: QIV08; U1111-1143-8433 (Other: WHO)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy; Influenza
Keywords: Quadrivalent Influenza Vaccine; Pregnancy Registry; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnancy Cases: Pregnant women exposed to Sanofi Pasteur's Quadrivalent Influenza Vaccine (QIV)
  Interventions: Biological: Quadrivalent Influenza Vaccine (QIV)

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine (QIV) — No Intervention as part of this protocol

SUMMARY:
The Sanofi Pasteur Quadrivalent Influenza Vaccine (QIV) Pregnancy Registry will be a prospectively recruited pregnancy surveillance program designed to collect and analyze information on vaccine exposures, pregnancy outcomes, and fetal and offspring outcomes.

DETAILED DESCRIPTION:
Pregnant women will be enrolled in the registry prospectively (after exposure to QIV in routine clinical settings but before knowledge of the pregnancy outcome). Women exposed to QIV with or without adverse events will be recorded in the Global Pharmacovigilance Database and medically reviewed. Pregnancy outcomes will be sought via questionnaires sent to the reporter at enrollment, estimated time of delivery, and six months after delivery. Descriptive statistical methods will be the primary approach for summarizing data.

No vaccine products will be provided or administered as part of this registry protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women will be enrolled in the registry prospectively (after exposure to Quadrivalent Influenza Vaccine (QIV) but before the conduct of any prenatal tests that could provide knowledge of the outcome of pregnancy). If the condition of the fetus has already been assessed through prenatal testing (e.g., targeted ultrasound, amniocentesis, etc.), such reports will be considered retrospective reports. Retrospective reports are also eligible for the registry but they will be analyzed separately from prospective reports.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women exposed to Sanofi Pasteur's Quadrivalent Influenza Vaccine (QIV)
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2013-08-16 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Number of cases and outcomes of pregnancies following exposure to QIV vaccine | Up to six years
  Data will be summarized using descriptive statistical methods and stratified by pregnancy outcome (spontaneous abortion, elective termination, fetal death/stillbirth, live birth) and timing of vaccine exposure. Infant outcomes include birth defects and physical and social development.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (5):
- United States (5):
  - San Diego, California
  - Albany, New York
  - Columbus, Ohio
  - Harrisburg, Pennsylvania
  - Nashville, Tennessee

REFERENCES:
- [Derived] Ledlie S, Gandhi-Banga S, Shrestha A, Mallett Moore T, Khromava A. Exposure to quadrivalent influenza vaccine during pregnancy: Results from a global pregnancy registry. Influenza Other Respir Viruses. 2022 Jan;16(1):90-100. doi: 10.1111/irv.12897. Epub 2021 Sep 14. PMID 34520127
- See also: Related Info — http://www.sanofipasteur.com
- See also: Related Info — http://www.sanofipasteurpregnancyregistry.com/